CLINICAL TRIAL: NCT06055413
Title: Remote Monitoring to Optimize Ventilatory Support in Children With Invasive Home Mechanical Ventilation
Brief Title: Home-based Optimization of Mechanical Ventilation in Children
Acronym: HOMVent4Kids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Carolyn Foster, Assistant Professor of Pediatrics, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-3600
Record Dates: First submitted 2023-09-14; First posted 2023-09-26 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Ventilator Weaning
Keywords: Children with medical complexity; Home mechanical ventilation; Long-term ventilation; Remote patient monitoring; Digital health
MeSH Terms: interventions — Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Patients receiving the intervention.
  Interventions: Other: Remote patient monitoring (RPM) bundle

INTERVENTIONS:
Other: Remote patient monitoring (RPM) bundle — Patient-families will be given a "remote patient monitoring (RPM) bundle" with tools to measure objective and subjective information about the child at home that are shared with the home ventilator provider team through an electronic dashboard. The tools include a device to measure carbon dioxide, a digital tablet, a digital weight scale, and a digital application that connects to the child's electronic health record. Each child will be assigned an individualized remote monitoring schedule (timing and data type) based on their indication for ventilation and ventilator regimen at enrollment.

SUMMARY:
Some children who are born very early or have other congenital conditions may develop severe, long-term lung problems that make them need to use a breathing machine to live at home. There are no studies that identify the best ways to monitor a home breathing machine or adjust its settings. Increasingly, healthcare systems are using information collected at home to make more informed decisions about a patient's healthcare treatment, which is called "remote patient monitoring". This study will ask whether using remote patient monitoring can provide more complete information to a child's team of doctors, nurses, and respiratory therapists to help a child's healthcare team and family make more informed decisions about a child's home ventilator care. The investigators are hypothesizing it can safely decrease the level of breathing support children need while also avoiding emergency and hospital care and supporting their growth, development, and participation in daily life.

DETAILED DESCRIPTION:
This is a single-arm, non-randomized, open-label trial using remote patient monitoring for chronic management of invasive home mechanical ventilation in children. The investigators hypothesize that integration of longitudinal physiologic data and patient reported outcome measures into routine clinical care over 4 months can optimize home mechanical ventilation use by 1) reducing the level home mechanical ventilation level of support, 2) improving patient and family quality of life, specifically participation in daily activities and patient's lung symptoms, and 3) improving family-reported shared decision-making and child's access to ventilator care. The investigators will also evaluate its usability within family life and provider workflows and assess early implementation outcomes.

ELIGIBILITY:
Family-Patient Inclusion criteria

* The patient uses invasive mechanical ventilation at home during any portion of the day at time of enrollment.
* The patient is 0 to 17 years old.
* The patient has at least one family caregiver (parent or other self-identified legal guardian) trained on home ventilator use who is willing to participate.
* The primary parental participant reads and speaks either English or Spanish.

Exclusion criteria

* The patient has progressive neuromuscular or other condition for which decreasing support during the day is not anticipated.
* The patient is already off of ventilation during the day while awake.
* The patient will turn 18 during participation.
* The patient has planned a transition of care to another institution or move during the planned study period after enrollment.
* The patient is in active hospice or similar end-of-life care at time of study enrollment.
* The patient is living in long-term institution, transitional facility, or not within a stable home setting during the study period.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Level of ventilator support | 4 months
  Liters/kg/day

SECONDARY OUTCOMES:
Cessation of awake positive pressure | 4 months
  Percentage of patients on any positive pressure ventilation during the day (per post discharge days)
Cessation of positive pressure | 4 months
  Percentage of patients on any positive pressure ventilation at any time (per post discharge days)
Ventilator management frequency | 4 months
  Number of ventilator management changes made per patient
Quality of life via participation | 4 months
  Two questions asking about to what extent the child's health issues interfered the child and the parent's with ability to engage in their usual activities. The questions are scored as 1, Not at all, 2, Slightly, 3, Moderately, 4, Quite a lot , 5, Extremely regarding how much the child's health affecting activity participation.
Lung symptom control | 4 months
  Parent report using bronchopulmonary dysplasia survey measure
Level of shared decision making | 4 months
  National Survey of Children's Health
  shared decision-making survey questions
Perceived access to ventilator care | 4 months
  Parent reported survey measure of their child's access to ventilator care
Child growth | 4 months
  Patient height and weight (absolute and Z scores)
Child healthcare utilization | 4 months
  Number of emergency department visits and hospitalizations.
Reach | 4 months
  To what degree potential patient participants participated, defined by comparing how many were approached versus participated.
Adoption | 4 months
  What percentage of eligible providers participated and what percentage of patients completed study.
Implementation | 4 months
  What was the rate of data collection and entry were completed by parents and reviewed by providers.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn C Foster, MD, MS, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foster C, Noreen P, Grage J, Kwon S, Hird-McCorry LP, Janus A, Davis MM, Goodman D, Laguna T. Predictors for invasive home mechanical ventilation duration in bronchopulmonary dysplasia. Pediatr Pulmonol. 2023 Jul;58(7):2085-2093. doi: 10.1002/ppul.26437. Epub 2023 Apr 28. PMID 37114844
- [Background] Foster CC, Kwon S, Shah AV, Hodgson CA, Hird-McCorry LP, Janus A, Jedraszko AM, Swanson P, Davis MM, Goodman DM, Laguna TA. At-home end-tidal carbon dioxide measurement in children with invasive home mechanical ventilation. Pediatr Pulmonol. 2022 Nov;57(11):2735-2744. doi: 10.1002/ppul.26092. Epub 2022 Aug 24. PMID 35959530
- See also: Foster Health Lab — https://sites.northwestern.edu/fosterhealthlab/
- See also: Primary Investigator — https://www.feinberg.northwestern.edu/faculty-profiles/az/profile.html?xid=38674